CLINICAL TRIAL: NCT02264444
Title: A Grading System for Laparoscopic Visualization and Predicting Factors That Affect Visualization Level During Laparoscopic Cholecystectomies: A Prospective, Single Group, Open Label Study
Brief Title: Establishing Visualization Grading Scale on LESS Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Hospital Tampa Bay Division (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Alexander Rosemurgy, Director HPB Surgery, GERD Center, Florida Hospital Tampa Bay Division
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 461326
Record Dates: First submitted 2014-10-01; First posted 2014-10-15 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Cholecystitis
Keywords: Cholecystectomy, visualization, single incision
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cholecystectomy visualization (Experimental): All patients will undergo a standard single site cholecystectomy and will have their operation recorded and scored for visualization.
  Interventions: Other: Cholecystectomy visualization

INTERVENTIONS:
Other: Cholecystectomy visualization — Patients undergo a standard removal of the gallbladder through a single incision at the umbilicus will have their operation recorded and graded according to a scale that is established for this study.

SUMMARY:
Essential to laparoscopic operations is adequate visualization. Unfortunately there is no grading system to assess the degree or quality of visualization. The primary objective of the project is to develop a laparoscopic visualization scoring system. We also intend to investigate the effects of neuromuscular blockade agents on visualization.

DETAILED DESCRIPTION:
Essential to laparoscopic operations is adequate visualization. Unfortunately there is no grading system to assess the degree or quality of visualization. There are many contributing factors that either assist or hinder the quality. Compared to open surgical procedures, laparoscopic surgical procedures (Laparo-endoscopic Single Site (LESS) and conventional multiport) are associated with less postoperative pain, a lower wound infection rate, shorter length of hospital stays and reduced incidence of late ventral hernia(1). Despite these well documented benefits of laparoscopic procedures, laparoscopy in certain patient populations can be challenging. Preoperative factors that contribute to technical difficulty in performance of laparoscopic procedures include male gender, android body habitus, and body mass index (BMI) greater than 30 kg/m2(2). Men often have an android body habitus, whereby the excess body fat concentrates within the peritoneal cavity, increases intra-abdominal pressure and thus reduces intraoperative laparoscopic visualization. Intra-abdominal pressure measured in morbidly obese patients is 2-3 times higher than in non-obese patients. In addition, android body habitus and high BMI are often associated with an enlarged left lobe of the liver. These factors can contribute to the degree of intraoperative technical difficulty and should be weighed in selection of appropriate patients to undergo laparoscopic procedures.

Particularly in the early period of the surgeon's learning curve, we suggest that selection criteria for laparoscopic procedures for the upper abdomen be limited to patients with a low BMI and no previous upper abdominal surgery. Although low BMI is a relatively good predictor of a less challenging laparoscopic procedure, a high BMI does not necessarily predict intraoperative technical difficulty. We predict that the best method to determine the technical difficulty of laparoscopic procedures is during intraoperative evaluation. For example, the primary limiting factor in determining the technical difficulty of laparoscopic Roux-en-Y gastric bypass (RYGBP) is the size and thickness of the left lobe of the liver. A massively enlarged left lobe of the liver obscures the laparoscopic view of the gastro-esophageal junction and angle of His, making the gastrojejunal anastomosis difficult to construct. Schwartz et al. support this concept when they found that a large liver was the primary reason for conversion from laparoscopic to open RYGBP in an analysis of 1,000 patients (2).

A laparoscopic operation consists of making small punctures into the peritoneum, through which, a camera and surgical instruments are subsequently inserted. The laparoscopically placed camera is the only view of the operative field. Since this point of view is constantly changing to meet the surgeon's needs during the operation, and because it is very different from the exoscopic view of the surgeon, the surgeon has to be very well trained to interpret the images through the laparoscopic view. For LESS operations, a deflectable tip laparoscope is utilized in aiding the surgeon for improved visibility and less clashing of instruments.

The laparoscopic view does not reveal, at one time, all the structures the surgeon needs to see in order to complete the surgical procedure with success. These structures can, for instance, be hidden behind the peritoneal wall (e.g., the ureter). This limitation cannot only lead to a less efficient operation, but can also lead to complications. Often such structures can be extracted from preoperative CT/MR images; however, the surgeon needs to interpret and fuse these images with the laparoscopic view. To alleviate this problem, we propose a laparoscopic visualization scoring system based on the intraoperative quality of images (3).

The impact of muscle relaxants on the isolated abdominal wall or diaphragmatic behavior and the absolute intra-abdominal volume are difficult to measure. Conversely, the inflated volume-pressure relationship of the abdominal cavity is easier to measure. A description of this volume-pressure relationship has not been identified in previous studies. Clinical data supports a positive linear correlation between the depth of neuromuscular blockade and abdominal wall and diaphragmatic relaxation and compliance (4). There is a very tangible and real effect of the neuromuscular blockade; this ultimately has a direct impact on the quality of visualization of the surgical field during a laparoscopic procedure (5). A constant neuromuscular block leads to preferable working conditions for the surgeon. The evoked muscle responses after neurostimulation can be registered by electromyography (EMG), mechanomyography (MMG) and acceleromyography (AMG). In principle, different peripheral nerves can be used for neurostimulation. The EMG records the electrical signal generated by the muscular action potential under its surface electrodes. The force of the thumb after stimulation can be registered by MMG. The AMG records the acceleration of the thumb after neurostimulation. The EMG, MMG and AMG system allows for observation of the measured signals quantity and quality (6).

We have identified other relevant factors that significantly affect the quality of visualization during different laparoscopic procedures including:

1. Clarity, focus and brightness:

   The laparoscope typically consists of an outer ring of optical fibers used to transmit light into the body, and an inner core of rod lenses that illuminate visual scene. This is then relayed back to the camera. Various different types of laparoscopes are available; they are specified in terms of overall length, number of rods, diameter and angle of view. Generally speaking, the wider the scope the brighter the resulting image. Lenses are available in the range of 1.9mm to 12mm, but sizes of 5mm and 10mm are the most common choices for pediatric and adult patients, respectively.
2. Breadth of intra-abdominal field and vertical space measured in centimeters:

   Breadth of intra-abdominal field and vertical space are factors directly related to pressure insufflation as well as the level of the neuromuscular blockade.
3. Distracting factors:

   This specific category of distracting factors includes:
   1. Blood: the presence, especially in large quantities, may prevent adequate visualization.
   2. Smoke: unipolar electrocautery and/or the bipolar Maryland forceps produce smoke when used. The rate of aspiration and evacuation also affect visualization.
   3. Adhesions: the presence of intra-abdominal adhesions, which hinders and prohibits proper identification of the anatomic structures.
   4. Sterile iodine impregnated covering sheet: its application presumably has a negative impact on abdominal wall and diaphragmatic compliance, and therefore, may obscure visualization.
   5. Intra-intestinal air: the presence of air inside the stomach, and small and large intestines adversely affects the size of the visual field. This can be prevented by an adequate preoperative bowel preparation and placement of an aspiration NG tube during anesthesia induction.
4. Patient's specific factors such as BMI value and body habitus:

   From our experience, a BMI under 26 allows for optimal field visualization. Conversely, a BMI greater than 26 negatively impacts the visual field. However, a recent study conducted by Camani et al. in 2010 showed that the laparoscopic approach in the various applications of gynecologic surgery is not significantly influenced by BMI in terms of surgical outcomes, laparotomy conversion rate, intraoperative and postoperative complication rate, and duration of hospital stay (4). We feel that visualization during operations involving the abdominal cavity are adversely affected by high amounts of adipose tissue, and therefore, a visualization scoring system will help support this theory.
5. Type of disorder (malignant vs. benign) that the laparoscopic procedure is undertaken for:

   Due to many pathologic factors such as the need for R0 resections, the discovery of more advanced disease than anticipated, the presence of adhesions or scar tissue from previous operations, laparoscopic procedures for malignant disorders may require a better visualization field than laparoscopic procedures undertaken for benign disorders.
6. Inadequate and/or poorly designed instruments:

   Most laparoscopic instrument development is technology-driven. This approach to instrument design does not always consider the ergonomics of the users, therefore leading to a user-unfriendly product (4, 5).
7. Technical difficulties:

   An intraoperative technical difficulty is defined as a significant deviation from the ordinary surgical procedure. All conversions to an open operation and iatrogenic bowel perforation during laparoscopic surgery are examples of technical difficulties. Many studies demonstrate that a technical difficulty during laparoscopic-assisted surgery jeopardizes both the intra-operative and postoperative patient safety.
8. Patient's body position during laparoscopic procedure:

A study led by Mulier, J et al. in 2010 demonstrated that the Trendelenburg position for lower abdominal surgery and reverse Trendelenburg with flexing of the legs at the hips for upper abdominal surgery effectively improved the workspace in obese patients, even with full muscle relaxation (6).

II. Objectives A.Primary Objective The primary objective is to develop a laparoscopic visualization scoring system.

B. Secondary Objectives

The secondary objectives are:

1. To determine how visualization is affected by various levels of pneumoperitoneum correlated with neuromuscular blockade.
2. Identify the factors that influence visualization, and determine how to manage these factors to optimize visualization.
3. Determine if there is a statistically significant correlation between different degrees of visualization and the following intraoperative time intervals:

   1. surgical incision to sterile wound dressing
   2. sterile wound dressing to extubation
   3. sterile wound dressing to patient exiting operating room
4. Determine if there is a statistically significant correlation between different degrees of visualization and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 18 years of age and older
* All patients deemed to have a clinical and surgical indication to undergo a LESS cholecystectomy

Exclusion Criteria:

1. Pregnancy
2. Breastfeeding
3. BMI>35
4. Serious comorbidities precluding a LESS cholecystectomy
5. Known or suspected neuromuscular disorders impairing neuromuscular function
6. Allergies to muscle relaxants, anesthetics or narcotics utilized for this study
7. A (family) history of malignant hyperthermia
8. A contraindication for neostigmine administration
9. Chronic opioid use
10. Prolonged QT syndrome
11. Creatinine >2.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Laparoscopic Visualization Score assessment | Start to end of LESS Cholecystectomy

SECONDARY OUTCOMES:
pneumoperitoneum volume | start to end of LESS cholecystectomy
factors influencing visualization | start to end of LESS cholecystectomy
Degrees of visualization | start to end of LESS cholecystectomy
  1. surgical incision to sterile wound dressing
  2. sterile wound dressing to extubation
  3. sterile wound dressing to patient exiting operating room
postoperative pain | every day until 7 days after LESS cholecystectomy

CONTACTS AND LOCATIONS:
Overall Officials: Alexander S. Rosemurgy, MD, Principal Investigator — Florida Hospital Tampa Bay Division
Locations (1):
- FloridaHTBD, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schrenk P, Woisetschlager R, Rieger R, Wayand WU. A diagnostic score to predict the difficulty of a laparoscopic cholecystectomy from preoperative variables. Surg Endosc. 1998 Feb;12(2):148-50. doi: 10.1007/s004649900616. PMID 9479730
- [Background] Nguyen NT, Longoria M, Gelfand DV, Sabio A, Wilson SE. Staged laparoscopic Roux-en-Y: a novel two-stage bariatric operation as an alternative in the super-obese with massively enlarged liver. Obes Surg. 2005 Aug;15(7):1077-81. doi: 10.1381/0960892054621062. PMID 16105411
- [Background] Stijn de Buck, Johan van Cleynenbreugel, Indra Geys, Thomas Koninckx, Philippe R Koninck, Paul Suetens. A System to Support Laparoscopic Surgery by Augmented Reality Visualization. Medical Image Computing and Computer-Assisted Intervention; 691-8, 2001.
- [Background] Camanni M, Bonino L, Delpiano EM, Migliaretti G, Berchialla P, Deltetto F. Laparoscopy and body mass index: feasibility and outcome in obese patients treated for gynecologic diseases. J Minim Invasive Gynecol. 2010 Sep-Oct;17(5):576-82. doi: 10.1016/j.jmig.2010.04.002. Epub 2010 Jul 8. PMID 20619751
- [Background] McDougall EM, Figenshau RS, Clayman RV, Monk TG, Smith DS. Laparoscopic pneumoperitoneum: impact of body habitus. J Laparoendosc Surg. 1994 Dec;4(6):385-91. doi: 10.1089/lps.1994.4.385. PMID 7881141
- [Background] Mulier JP, Dillemans B, Van Cauwenberge S. Impact of the patient's body position on the intraabdominal workspace during laparoscopic surgery. Surg Endosc. 2010 Jun;24(6):1398-402. doi: 10.1007/s00464-009-0785-8. Epub 2010 Jan 7. PMID 20054583
- [Background] Simanski , R. Kahler, B. Pohl, R. Hofmockel, R. Friedrich, B. P. Lampe Measurement and control of neuromuscular blockade and depth of anaesthesia. Proceedings of the European Control Conference, Cambridge/UK. 2003.